CLINICAL TRIAL: NCT00541138
Title: A Pilot Study of Tamoxifen, Carboplatin and Topotecan in the Treatment of Recurrent or Refractory Primary Brain or Spinal Cord Tumors or Metastatic Epithelial Cancers With Central Nervous System Metastases
Brief Title: Tamoxifen, Carboplatin, and Topotecan in Treating Patients With CNS Metastases or Recurrent Brain or Spinal Cord Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02191; P30CA033572 (NIH); CHNMC-02191; CDR0000570253 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: tumors metastatic to brain; recurrent adult brain tumor; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; adult pilocytic astrocytoma; adult pineal gland astrocytoma; adult subependymal giant cell astrocytoma; adult brain stem glioma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic oligodendroglioma; adult oligodendroglioma; unspecified adult solid tumor, protocol specific; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Astrocytoma; Glioblastoma; Gliosarcoma; Ependymoma; Glioma, Subependymal; Oligodendroglioma; Glioma | interventions — Carboplatin; Tamoxifen; Topotecan

INTERVENTIONS:
Drug: carboplatin — CBDCA AUC=3
Drug: tamoxifen citrate — Tamoxifen 100mg bid
Drug: topotecan hydrochloride — Topotecan 0.75 g/m2/d
Other: pharmacological study — Start of tx, hours 24,28 and 72 during Topotecan infusion, and hours 1,2,4 and 6 after end of Topotecan infusion.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and topotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Tamoxifen may help carboplatin work better by making tumor cells more sensitive to the drug.

PURPOSE: This phase II trial is studying the side effects of giving carboplatin and topotecan together with tamoxifen and to see how well it works in treating patients with central nervous system metastases or recurrent brain or spinal cord tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the systemic and CNS response rates and progression-free and overall survival of patients with epithelial cancer and brain metastases treated with tamoxifen citrate, topotecan hydrochloride, and carboplatin.
* To evaluate the response rates, progression-free survival, and overall survival of patients with recurrent primary glial tumors treated with this regimen.
* To further assess the toxicity of these drugs in these patients.
* To further evaluate the pharmacokinetics of topotecan hydrochloride and tamoxifen citrate using paired specimens of cerebrospinal fluid and plasma from these patients.

OUTLINE: Patients are stratified by disease type (epithelial CNS metastases vs recurrent glial tumors).

Patients receive topotecan IV on days 1-3 (72 hours), carboplatin IV over 30 minutes on day 4, and oral tamoxifen twice daily on days 1-7. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) may be treated for 2 additional courses after documentation of CR.

Patients undergo blood sample collection at baseline and then periodically after the first dose of topotecan to obtain plasma pharmacokinetic (PK) measurements of topotecan and tamoxifen. Some patients may also undergo cerebrospinal fluid (CSF) collection to assess peak CSF levels of topotecan and tamoxifen during course 1.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Epithelial neoplasms metastatic to the central nervous system

    * Recurrent or refractory to prior chemotherapeutic or radiotherapeutic regimens or for which no standard chemotherapy or whole brain radiotherapy regimens exist
    * Stage IV disease
  * Recurrent glial tumors (brain or spinal cord)
* Received prior whole brain radiotherapy or stereotactic radiotherapy OR refused radiotherapy

  * Patients with CNS metastases previously treated with radiotherapy are eligible, provided persistent or progressive CNS metastases are documented by MRI eight weeks after the end of radiotherapy
  * Patients with glial tumors must show progressive disease by MRI after prior radiotherapy
* Measurable disease in the brain/leptomeninges of the brain or spinal cord with baseline documentation within 4 weeks of study entry

  * Must have ≥ 1 lesion that is ≥ 1 cm on MRI scan
* Ineligible for or has refused participation in higher priority institutional protocols

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Life expectancy ≥ 2 months
* Creatinine ≤ 1.5 mg/dL
* WBC 4,000/mm³ OR ANC ≥ 2,000/mm³
* Platelet count ≥ 150,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST < 2 times upper limit of normal
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No nonmalignant concurrent illness (e.g., cardiovascular or pulmonary) that is either poorly controlled with currently available treatment or of such severity to preclude study entry
* No severe infection
* Patients who are ineligible for lumbar puncture are allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy, immunotherapy, or chemotherapy OR recovered from expected side effects of prior therapy
* No patients who are recovering from major surgery
* No concurrent radiotherapy
* Concurrent steroid or anticonvulsant therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Toxicity profile as assessed by NCI CTC v2.0 | All patients who complete one course of therapy and are followed a minimum of 3 weeks after completion of first course of therapy
Response rate in patients with recurrent glial tumors as assessed by RECIST criteria | All patients who complete at least one cycle of treatment
Response rate in patients with epithelial CNS metastases as assessed by RECIST criteria | All patients who complete at least one cycle of treatment
Reason for going off-study | Reported for all eligible patients
Progression | Reported for all eligible patients
Survival | Reported for all eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Morgan, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States